CLINICAL TRIAL: NCT03433560
Title: An Observational, Prospective, Open Label, Multicenter Study to Evaluate the Safety and Efficacy of Pegfilgrastim (Neulasta®) as Secondary Prophylaxis to Decrease the Incidence of Febrile Neutropenia in Korean Female Patients With Breast Cancer.
Brief Title: An Observational Study to Evaluate the Safety and Efficacy of Pegfilgrastim (Neulasta®)
Status: Completed | Type: Observational
Sponsor: Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: KKKR-Neulasta OS-01
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Female; Breast Neoplasm Female
Keywords: febrile neutropenia; neutropenia
MeSH Terms: conditions — Febrile Neutropenia; Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to evaluate real-world safety and efficacy of pegfilgrastim (Neulasta) administered as secondary prophylaxis in Korean female patients with breast cancer receiving chemotherapy regimens recently covered under national health insurance. This is a prospective, observational, open-label trial with a target enrollment of 1400 subjects.

Primary endpoint The primary aim of this study is to determine the incidence of febrile neutropenia.

Secondary endpoint Major secondary endpoint include a) Incidence of bone pain, b) All adverse events, c) Percentage of patients with RDI (relative dose intensity) ≥ 85%

ELIGIBILITY:
Inclusion Criteria:

* ≥ 19 years old, and ≤ 64 years old, and
* Female patients with breast cancer receiving chemotherapy recently covered under national health insurance (only chemotherapy regimens in the table below), and
* Patients with neutropenic events (febrile neutropenia or grade 4 neutropenia) in any previous cycle that did not use G-CSF for the prevention of neutropenia

Exclusion Criteria:

Patients with any of the followings are excluded.

* Patients with a history of allergic reactions to E-coli derived proteins, human granulocyte colony-stimulating factors such as pegfilgrastim or filgrastim
* Uses for off-label indications such as chronic myelogenous leukemia, myelodysplastic syndrome

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Please refer to the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of febrile neutropenia after secondary prophylaxis with pegfilgrastim | From the cycle of chemotherapy before administration of next cycle of chemotherapy (approximately 3weeks)

SECONDARY OUTCOMES:
The incidence of bone pain, or percentage of patients with relative dose intensity (RDI) or all adverse events as assessed by CTCAE | During the study period (~ 1months follow-up)

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Bucheon Soonchunhyang University Hospital, Bucheon-si, Kyounggi
  - Pusan National University Yangsan Hospital, Yangsan, Kyoungsang